CLINICAL TRIAL: NCT05784428
Title: Single vs. Multiple Fraction Non-Inferiority Trial of Stereotactic Ablative Radiotherapy for the Comprehensive Treatment of Oligo-metastases/Progression: SIMPLIFY-SABR-COMET
Brief Title: Single vs. Multiple Fraction Trial of Stereotactic Ablative Radiotherapy for Comprehensive Treatment of Oligometastases/Progression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Olson (Other)
Collaborators: London Regional Cancer Program, Canada (Other); Tom Baker Cancer Centre (Other); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor-Investigator, Robert Olson, Radiation Oncologist, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SIMPLIFY-SABR-COMET
Record Dates: First submitted 2023-02-28; First posted 2023-03-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Oligometastatic Disease; Oligoprogression; Toxicity Due to Radiotherapy; Quality of Life

STUDY DESIGN:
Intervention Model Description: This study is a phase III multicentre randomized trial. All participants will be randomized in a 1:1 ratio between multiple fraction SABR (Arm 1) vs. single fraction SABR (Arm 2). Patients will be stratified by systemic therapy within the last 2 weeks (yes/no); number of sites to be treated (1 vs. multiple) and SABR to the abdominal/pelvic site (yes/no).
  BC Cancer sites will also participate in the second randomization. Participants will be randomized in a 1:1 ratio to QoL reporting alone via FACT-G and EQ-5D-5L (Arm A) vs. QoL reporting and patient-reported outcome (PRO) symptom screen with healthcare provider intervention (Arm B). Patients will be further stratified by the criteria for the 1st randomization as as well as sex.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Multiple fraction SABR (Arm 1) (Active Comparator): Participants randomized to this arm will receive multiple fraction SABR
  Interventions: Radiation: Multiple fraction SABR
- Single fraction SABR (Arm 2) (Experimental): Participants randomized to this arm will receive single fraction SABR
  Interventions: Radiation: Single fraction SABR
- Patient-reported outcome (PRO) collection : QoL reporting alone (Arm A) (Active Comparator): Participants will complete the EuroQoL-5Dimensions-5levels (EQ-5D-5L) and Functional Assessment of Cancer Therapy-General (FACT-G) prior to each scheduled follow-up (FU).
  Interventions: Other: QoL reporting alone
- QoL reporting and healthcare provider (HCP) intervention guided by symptom screen (Arm B) (Experimental): * Patients complete EQ-5D-5L and FACT-G prior to each scheduled FU
  * Patient complete online adaptive symptom screen with HCP intervention, prior to each scheduled appointment
  Interventions: Other: QoL reporting, symptom screen and healthcare provider intervention

INTERVENTIONS:
Radiation: Single fraction SABR — Participants randomized to this arm will receive SF SABR
  Treatment recommendations are as follows:
  Lung: Greater than 2 cm from mediastinum or brachial plexus or if mandatory OAR constraints are met: 30 Gy in 1 fraction
  Lung: Within 2 cm of mediastinum or brachial plexus 20 Gy in 1 fraction
  Bone, Spine, Adrenal, lymph node/soft tissue: 20 Gy in 1 fraction
  Liver: 30 Gy in 1 fraction
  Brain: dose as per institutional policy
  Arms: Single fraction SABR (Arm 2)
Radiation: Multiple fraction SABR — Participants randomized to this arm will receive MF SABR:
  Dose/Fractionation are as follows:
  Lung: Greater than 2 cm from mediastinum or brachial plexus or if mandatory organ-at-risk (OAR) constraints are met: 48 Gy in 4 fractions (12 Gy/#), 54 Gy in 3 fractions (18 Gy/#), daily or every second day
  Lung: Within 2 cm of mediastinum or brachial plexus 60 Gy in 8 fractions (7.5 Gy/#), 50 Gy in 5 fractions (10 Gy/#), daily
  Bone: Any bone except spine: 35 Gy in 5 fractions (7 Gy/#), daily
  Liver: 54 Gy in 3 fractions (18 Gy/#) or 5 fractions (10.8 Gy/#), daily or every second day
  Spine: 24 Gy in 2 fractions (12 Gy/#) or 35 Gy in 5 fractions (7 Gy/#), daily
  Adrenal: 40 Gy in 5 fractions (8 Gy/#) or 35 Gy in 5 fractions (7 Gy/#), daily
  Lymph node/soft tissue: 40 Gy in 5 fractions (8 Gy/#) or 35 Gy in 5 fractions (7 Gy/#), daily
  Brain - dose per institutional policy for stereotactic lesions (no whole brain RT).
  Arms: Multiple fraction SABR (Arm 1)
Other: QoL reporting alone — Participants randomized to this arm will complete the EQ-5D-5L and FACT-G at baseline and each follow-up visit
  Arms: Patient-reported outcome (PRO) collection : QoL reporting alone (Arm A)
Other: QoL reporting, symptom screen and healthcare provider intervention — Participants randomized to this arm will complete the FACT,G, EQ-5D-5L, radiation-symptom screen and receive healthcare provider-guided intervention based on their symptom reports.
  Arms: QoL reporting and healthcare provider (HCP) intervention guided by symptom screen (Arm B)

SUMMARY:
Stereotactic Ablative Radiotherapy (SABR) is a modern RT technique that delivers high doses of radiation to small tumor targets using highly conformal techniques, while trying to avoid healthy tissues and organs. However, SABR treatment requires increased planning, treatment time, cost and potential for higher toxicity due to the higher dose. The purpose of this study is to compare single fraction (SF) SABR vs. multiple fraction (MF) SABR in regards to toxicities, progression-free survival, quality of life (QoL), and cost-effectiveness. In a subset of patients, we will also compare patient QoL, hospitalization rates, and cost-effectiveness between patients who complete QoL questionnaires, record symptoms and receive healthcare provider-guided intervention vs. patients who complete QoL questionnaires only.

DETAILED DESCRIPTION:
Radiation can be delivered in multiple fractions, or doses, and can take up to several weeks or months of treatment depending on the type of cancer. Radiation can also be offered in a single fraction. Both techniques have evidence for use in clinical care. Multiple fraction is offered to reduce the amount of radiation given at a single time that could reduce late toxicities. However, single fraction radiotherapy is more cost-effective and saves patient time. With this trial, we will compare single fraction vs. multiple fraction in regards to their impact on toxicity, progression-free survival: time from randomization to disease progression at any site or death, lesional control rate: lesion size post-SABR, quality of life and cost-effectiveness.

In a subset of sites, we will also investigate the impact of healthcare-provider guided intervention on quality of life. Questionnaires capture various symptoms such as pain, fatigue and information relating to physical, social, and mental wellbeing. This information can help shed light on patient experience and provide a better understanding of the effects of radiation therapy. In this trial, we will compare quality of life questionnaire completion, symptom reporting and healthcare-provider guided intervention vs. quality of life questionnaire completion alone, in regards to patient quality of life. Hospitalization rates and frequency of emergency department visits will also be investigated.

Sample size: The total sample size of 598 for this trial was calculated based on the primary endpoint of toxicity for the single vs. multiple fraction SABR randomization. Calculations were performed based on the results of the SABR-5 trial and our clinical judgement.

Quality Assurance: Radiation treatments are based on the current phase III SABR-COMET-3 trial and as per recent clinical evidence. All treatments will be planned as per protocol including computed tomography (CT) simulation, organs at risk contouring and undergo a quality assurance process.

For the subset of sites involved in the second randomization, training will be provided to patients on the use of Noona, a patient-reported outcome platform.

ELIGIBILITY:
Inclusion Criteria:

* 1-5 current oligometastatic or oligo-progressive lesions
* Age 18 years or older
* Able to provide informed consent
* Able to complete electronic entry of patient reported outcomes and questionnaires independently or with assistance from a caregiver/family/friend/research staff using electronic methods after providing consent to email use.
* Life expectancy > 6 months
* Histologically confirmed malignancy with metastatic disease detected on imaging. Biopsy of metastasis is preferred, but not required.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Controlled primary tumor: defined as at least 3 months since original tumor treated radically, with no progression at primary site (can be considered controlled if no evidence of the primary tumour on imaging [e.g. primary unknown])
* A history and physical examination, including ECOG performance status, performed within 6 weeks prior to enrollment
* Patient has had a CT chest, abdomen and pelvis or PET-CT within 10 weeks prior to enrollment, and within 13 weeks prior to treatment
* Patient has had a nuclear bone scan (if no positron emission tomography-computed tomography [PET-CT]) within 10 weeks prior to enrollment, and within 13 weeks prior to treatment
* Patient has had CT or MRI brain imaging if primary has a propensity for central nervous system metastases within 10 weeks prior to enrollment, and within 13 weeks prior to treatment.
* For patients with known spine metastases, patient has had MRI spine imaging within 10 weeks prior to enrollment, and with 13 weeks prior to treatment.
* If solitary lung nodule for which biopsy is unsuccessful or not possible, patient has had an FDG (fluorodeoxyglucose) PET scan or CT (chest, abdomen, pelvis) and bone scan within 10 weeks prior to enrollment, and within 13 weeks prior to treatment
* If colorectal primary with rising Carcinoembryonic antigen (CEA), but equivocal imaging, patient has had an FDG PET scan within 10 weeks prior to enrollment, and within 13 weeks prior to treatment
* Patient is judged able to:

  * Maintain a stable position during therapy
  * Tolerate immobilization device(s) that may be required to deliver SABR safely
* Negative pregnancy test for People of Child-Bearing Potential (POCBP) within 4 weeks of RT start date

Waivers to inclusion criteria will NOT be allowed.

Exclusion Criteria:

* Uncontrolled concurrent malignant cancer
* Lesion in femoral bone requiring surgical fixation
* No chemotherapy agents (cytotoxic, or molecularly targeted agents) will be used within the period of time commencing 1 week prior to radiation, lasting until 1 week after the last fraction. See section 5.3.3 regarding this criterion.
* Serious medical comorbidities precluding radiotherapy. These include interstitial lung disease in patients requiring thoracic radiation, Crohn's disease in patients where the gastrointestinal (GI) tract will receive radiotherapy, and connective tissue disorders such as lupus or scleroderma.
* Substantial overlap with a previously treated radiation volume. Prior radiotherapy in general is allowed, as long as the composite plan meets dose constraints herein. For patients treated with radiation previously, similar biological effective dose calculations should be used to equate previous doses to the tolerance doses listed below. All such cases should be discussed with the local and study principal investigators (PIs).
* Current malignant pleural effusion
* Liver metastases located in the "Biliary no fly zone" defined for this trial as common biliary track, cystic duct and distal branches (1 cm) + 5 mm.
* Inability to treat all sites of oligometastatic or oligoprogressive disease
* Maximum size of 5 cm for lesions outside the brain, except:

  * Bone metastases over 5 cm may be included, if in the opinion of the local PI it can be treated safely (e.g. rib, scapula, pelvis)
  * Any brain metastasis > 3.5 cm in size or a total volume of brain metastases greater than 30 cc is excluded
* Clinical or radiologic evidence of spinal cord compression. Patients can be eligible if surgical resection has been performed
* Patients with spine instability as judged by a Spinal Instability Neoplastic Score (SINS) of >12
* Dominant brain metastasis requiring surgical decompression
* Surgical resection of all metastases (i.e. no lesion available to be treated with SABR)
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2035-04-30 (Estimated); Study Completion 2035-05-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | At 6 weeks, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Occurrences and changes in grade 3 or higher adverse events related to treatment, according to CTCAE v5.0
Change in patient-reported quality of life | At 6 weeks, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  As measured by the EQ-5D-5L. This questionnaire provides measures for mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It also includes a numbered scale from 0 to 100 where 100 means the best health one can imagine, and 0 means the worst health one can imagine.

SECONDARY OUTCOMES:
Lesional control rate | At 6 weeks, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Rate is determined based on lesion size post-SABR using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Progression-free survival | At 6 weeks, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Time from randomization to disease progression at any site or death
Overall survival | Approximately at the end of year 5 of follow-up, at study completion
  Time from randomization to death from any cause (exploratory)
Resource utilization | At 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Assessed via patient- and provider-reported hospitalization rates, frequency of emergency department visits, number of patients with systemic or radiation therapy post SABR treatment on trial

CONTACTS AND LOCATIONS:
Overall Officials: Robert Olson, MD, MSc, FRCPC, Principal Investigator — BC Cancer - Prince George
Locations (13):
- Canada (6):
  - BC Cancer, Kelowna, British Columbia
  - BC Cancer, Prince George, British Columbia
  - BC Cancer, Surrey, British Columbia
  - BC Cancer, Vancouver, British Columbia
  - BC Cancer - Victoria, Victoria, British Columbia
  - Princess Margaret Cancer Centre | University Health Network, Toronto, Ontario
- Ireland (7):
  - University Hospital Galway, Galway, Connacht
  - St. Luke's Radiation Oncology Network, Dublin, Dublin
  - Mater Private Hospital, Dublin, Leinster
  - Beacon Hospital, Dublin, Leinster
  - Cork University Hospital, Cork, Munster
  - Bon Secours Radiotherapy Cork in Partnership with UPMC Hillman Cancer Centre, Cork, Munster
  - UPMC Whitfield Hospital - Waterford, Waterford, Munster

REFERENCES:
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Patel PH, Palma D, McDonald F, Tree AC. The Dandelion Dilemma Revisited for Oligoprogression: Treat the Whole Lawn or Weed Selectively? Clin Oncol (R Coll Radiol). 2019 Dec;31(12):824-833. doi: 10.1016/j.clon.2019.05.015. Epub 2019 Jun 8. PMID 31182289
- [Background] Nguyen TK, Chin L, Sahgal A, Dagan R, Eppinga W, Guckenberger M, Kim JH, Lo SS, Redmond KJ, Siva S, Stish BJ, Chan R, Lawrence L, Lau A, Tseng CL. International Multi-institutional Patterns of Contouring Practice and Clinical Target Volume Recommendations for Stereotactic Body Radiation Therapy for Non-Spine Bone Metastases. Int J Radiat Oncol Biol Phys. 2022 Feb 1;112(2):351-360. doi: 10.1016/j.ijrobp.2021.09.004. Epub 2021 Sep 9. PMID 34509549
- [Background] Cox BW, Spratt DE, Lovelock M, Bilsky MH, Lis E, Ryu S, Sheehan J, Gerszten PC, Chang E, Gibbs I, Soltys S, Sahgal A, Deasy J, Flickinger J, Quader M, Mindea S, Yamada Y. International Spine Radiosurgery Consortium consensus guidelines for target volume definition in spinal stereotactic radiosurgery. Int J Radiat Oncol Biol Phys. 2012 Aug 1;83(5):e597-605. doi: 10.1016/j.ijrobp.2012.03.009. Epub 2012 May 19. PMID 22608954
- [Background] Redmond KJ, Robertson S, Lo SS, Soltys SG, Ryu S, McNutt T, Chao ST, Yamada Y, Ghia A, Chang EL, Sheehan J, Sahgal A. Consensus Contouring Guidelines for Postoperative Stereotactic Body Radiation Therapy for Metastatic Solid Tumor Malignancies to the Spine. Int J Radiat Oncol Biol Phys. 2017 Jan 1;97(1):64-74. doi: 10.1016/j.ijrobp.2016.09.014. Epub 2016 Sep 17. PMID 27843035
- [Background] Dunne EM, Sahgal A, Lo SS, Bergman A, Kosztyla R, Dea N, Chang EL, Chang UK, Chao ST, Faruqi S, Ghia AJ, Redmond KJ, Soltys SG, Liu MC. International consensus recommendations for target volume delineation specific to sacral metastases and spinal stereotactic body radiation therapy (SBRT). Radiother Oncol. 2020 Apr;145:21-29. doi: 10.1016/j.radonc.2019.11.026. Epub 2019 Dec 23. PMID 31874346
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Common Terminology Criteria for Adverse Events (CTCAE) Common Terminology Criteria for Adverse Events (CTCAE) v5.0. 2017
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Basch E, Reeve BB, Mitchell SA, Clauser SB, Minasian LM, Dueck AC, Mendoza TR, Hay J, Atkinson TM, Abernethy AP, Bruner DW, Cleeland CS, Sloan JA, Chilukuri R, Baumgartner P, Denicoff A, St Germain D, O'Mara AM, Chen A, Kelaghan J, Bennett AV, Sit L, Rogak L, Barz A, Paul DB, Schrag D. Development of the National Cancer Institute's patient-reported outcomes version of the common terminology criteria for adverse events (PRO-CTCAE). J Natl Cancer Inst. 2014 Sep 29;106(9):dju244. doi: 10.1093/jnci/dju244. Print 2014 Sep. PMID 25265940
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Olson R, Mathews L, Liu M, Schellenberg D, Mou B, Berrang T, Harrow S, Correa RJM, Bhat V, Pai H, Mohamed I, Miller S, Schneiders F, Laba J, Wilke D, Senthi S, Louie AV, Swaminath A, Chalmers A, Gaede S, Warner A, de Gruijl TD, Allan A, Palma DA. Stereotactic ablative radiotherapy for the comprehensive treatment of 1-3 Oligometastatic tumors (SABR-COMET-3): study protocol for a randomized phase III trial. BMC Cancer. 2020 May 5;20(1):380. doi: 10.1186/s12885-020-06876-4. PMID 32370765
- [Derived] Olson R, Abraham H, Leclerc C, Benny A, Baker S, Matthews Q, Chng N, Bergman A, Mou B, Dunne EM, Schellenberg D, Jiang W, Chan E, Atrchian S, Lefresne S, Carolan H, Valev B, Tyldesley S, Bang A, Berrang T, Clark H, Hsu F, Louie AV, Warner A, Palma DA, Howell D, Barry A, Dawson L, Grendarova P, Walker D, Sinha R, Tsai J, Bahig H, Thibault I, Koul R, Senthi S, Phillips I, Grose D, Kelly P, Armstrong J, McDermott R, Johnstone C, Vasan S, Aherne N, Harrow S, Liu M. Single vs. multiple fraction non-inferiority trial of stereotactic ablative radiotherapy for the comprehensive treatment of oligo-metastases/progression: SIMPLIFY-SABR-COMET. BMC Cancer. 2024 Feb 3;24(1):171. doi: 10.1186/s12885-024-11905-7. PMID 38310262